CLINICAL TRIAL: NCT01762852
Title: BEL114674: A 2 Year Study of Efficacy and Safety of Intravenous Belimumab Versus Placebo in Subjects With Idiopathic Membranous Nephropathy
Brief Title: Efficacy and Safety Study of Intravenous Belimumab Versus Placebo in Subjects With Idiopathic Membranous Nephropathy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn due to difficulties in to recruiting due to competing studies, changing treatment practices, unavailability of eligible study population
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 114674
Record Dates: First submitted 2013-01-04; First posted 2013-01-08 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Glomerulonephritis, Membranous
Keywords: Benlysta; efficacy; proteinuria; Idiopathic membranous nephropathy; GSK1550188; anti-phospholipase A2 receptor antibodies; safety; placebo; BLyS; belimumab; Lymphostat-B; membrane attack complex
MeSH Terms: conditions — Glomerulonephritis, Membranous; Proteinuria | interventions — belimumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Belimumab Arm (Experimental): Subjects will receive belimumab 10 mg/kg intravenous infusion [will last for 1 hour (hr)] on Day 0, Week 2, Week 4, then every 4 weeks for up to 100 weeks with frequency adjusted for subjects with >1000 mg/mmol uPCR (>10 g/24 hrs). All subjects will receive background supportive therapy throughout the study.
  Interventions: Drug: Belimumab 10 mg
- Placebo Arm (Placebo Comparator): Intravenous infusion (will last for 1 hr) on Day 0, Week 2, Week 4, then every 4 weeks for up to 100 weeks with frequency adjusted for subjects with >1000 mg/mmol uPCR (>10 g/24 hrs). All subjects will receive background supportive therapy throughout the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Belimumab 10 mg — Belimumab is Lyophilised powder for reconstitution in 4.8 mL sterile water for injection (SWFI) and diluted in normal saline (250 mL). 400 mg per vial plus excipients (citric acid/sodium citrate/sucrose/polysorbate). Belimumab 10 mg/kg intravenous infusion (will last for 1 hr) on Day 0, Week 2, Week 4, then every 4 weeks for up to 100 weeks
  Arms: Belimumab Arm
Drug: Placebo — Normal saline solution (sodium chloride 154 mmol/L). Intravenous infusion (will last for 1 hr) on Day 0, Week 2, Week 4, then every 4 weeks for up to 100 weeks
  Arms: Placebo Arm

SUMMARY:
The main clinical study will be a randomized, double-blind, placebo-controlled, long term study involving a 100 week treatment period. The purpose of this study is to test for superiority of treatment with belimumab 10 mg/kg plus supportive therapy compared to placebo plus supportive therapy in idiopathic membranous nephropathy (IMN). The purpose of this study is also to investigate the effect of initiating earlier treatment with belimumab compared to delayed treatment with current immunosuppressive treatment regimens. The study will also determine the pharmacokinetic (PK) profile of belimumab and further explore the mechanism of action of Belimumab as well as effects on quality of life. All subjects (on either active treatment or placebo) will receive background supportive therapy throughout the main clinical study, which includes angiotensin-converting enzyme inhibitors (ACEi) and/or angiotensin receptor blockers (ARBs) unless contraindicated and may include statins, diuretics, dietary salt restriction but excludes immunosuppressants (except low dose corticosteroids). Screening will be done within 5 to 2 weeks before the first scheduled dose of study treatment. A total of 94 evaluable subjects will be randomized in a 1:1 ratio such that 47 subjects receive intravenous belimumab 10 mg/kg and 47 receive intravenous placebo. Subjects will be dosed on Days 0, 14, 28 and then every 4 weeks through to, and including, Week 100, resulting in a total of 27 doses (giving 104 weeks of drug exposure). The dosing frequency will be adjusted to every 2 weeks if the subject's proteinuria as assessed by urinary protein creatinine ratio (PCR) is greater than 1000mg/mmol (greater than 10 g/24 h), to compensate for loss of belimumab in the urine. Subjects who are withdrawn from study treatment at any time during the study, eg for rescue therapy, will participate in follow-up visits every 12 weeks up to week 104. A subject will be regarded as having completed the main clinical study if they complete all phases of the main clinical study (screening, treatment period, 4 week and 16 week post last dose short term safety follow-up). Subjects who complete the main clinical study will therefore participate in the main clinical study for approximately 28 months. After the main clinical study, there will be a 5 year (long term) follow-up phase to assess long term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age & Gender: Male or female between 18 and 75 years of age inclusive, at the time of signing the informed consent.
* Histological diagnosis: Have clinical diagnosis of IMN, as verified by biopsy (either by light microscope with immuno-fluorescence, or by electron microscope) in the last 3 years (biopsy results [and slides where possible] should be available for independent evaluation). For patients with relapsed disease, a biopsy should be available within the preceding 7 years.
* Proteinuria: Have clinically active disease (nephrotic range proteinuria) for at least 3 months prior to screening and no improvement (<30% reduction), despite supportive therapy (which must include maximal tolerated doses of ACE inhibitor or ARB unless contraindicated, and may include statins, diuretics, dietary salt restriction). During screening proteinuria must be >400 mg/mmol by uPCR (or >4.0 g per 24 hrs) as measured from a 24 hrs urine collection and/or spot urine sample (early morning where possible) on 2 occasions at least 7 days apart.
* Proteinuria in patients with relapsed disease: Patients who previously achieved proteinuria <2 g per 24h for at least 6 months and have subsequently relapsed with proteinuria levels as documented above, may be eligible providing recurrence has been within the previous 3 years and patient is known to be anti-PLA2R positive.
* Female Subject is eligible to participate if she is not pregnant or nursing; is non-childbearing potential. Females of child-bearing potential must agree to use one of the approved contraception methods for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimise the risk of pregnancy at that point. Female subjects must agree to use contraception until 16 weeks after the last dose.
* French subjects: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.
* Inclusion Criteria for Long Term Follow-up: Subjects who have signed informed consent for the Long Term Follow-up and have completed 2 years study treatment and the 16 week follow-up visit, or who have withdrawn early from study treatment but completed the Week 104 Withdrawn visit.

Exclusion Criteria:

* Non-Idiopathic MN or other condition affecting the kidney: If the diagnosis of MN is secondary to other conditions, or the subject has renal impairment from a condition that is not MN. Causes of secondary MN include (but are not limited to) Immune diseases (Systemic lupus erythematosus, diabetes mellitus; rheumatoid arthritis, Hashimoto's disease, Grave's disease, mixed connective tissue disease, Sjogren's syndrome, primary biliary cirrhosis, bullous pemphigoid, small bowel enteropathy syndrome, dermatitis herpetiformis, ankylosing spondylitis, graft-versus-host-disease, Guillain-Barre syndrome); or Infectious or parasitic diseases (Hepatitis B; Hepatitis C, syphilis, filariasis, hydatid disease, schistosomiasis, malaria, leprosy); or Drugs and toxins (Gold, penicillamine, non-steroidal anti-inflammatory agents, mercury, captopril, formaldehyde, hydrocarbons, bucillamine); or Miscellaneous(Tumors excluded with reasonable diligence, renal transplantation, sarcoidosis, sickle cell disease, Kimura disease, angiofollicular lymph node hyperplasia).
* Anti-PLA2R autoantibody: Patients known to be negative for anti-PLA2R autoantibody.
* Severely reduced or deteriorating kidney function: An eGFR at screening <40 mL/min/1.73m^2 (as determined by 4 variable version MDRD equation) or kidney function not stable (as defined by >15% decrease in eGFR in 3 months before screening unless due to medication change).
* Blood Pressure: Uncontrolled hypertension defined as blood pressure (BP) >150/90 mmHg (treatment target <=140/80)
* Prior Therapy: Have received treatment with the following therapies at the times specified prior to Day 0: Therapy - B-cell targeted therapy except rituximab (e.g., other anti- CD20 agents, anti-CD22 [epratuzumab], anti-CD52 [alemtuzumab], BLyS-receptor fusion protein [BR3], TACI Fc, or belimumab), Time period: anytime; Therapy: Rituximab (subjects with rituximab treatment between 1 and 2 years prior to Day 0 are eligible if there is documented evidence of B-cell repopulation to >50% of pre-treatment levels), Period: 2 years; Therapy: Abatacept and any other biologic investigational agent other than B cell targeted therapy (i.e. not approved for sale in the country in which it is being used), Time Period: 364 days; Therapy: Cyclophosphamide or chlorambucil 3 or more courses of systemic corticosteroids for concomitant conditions (e.g., asthma, atopic dermatitis). (Topical or inhaled steroids are permitted.), Time Period: 180 days; Therapy: Anti-tumour necrosis factor (TNF) or anti-IL-6 therapy (e.g. adalimumab, etanercept, infliximab, tocilizumab). Interleukin-1 receptor antagonists (e.g. anakinra). Other immunosuppressive/immunomodulatory agents (e.g azathioprine, 6-mercaptopurine, mycophenolate mofetil (PO)/ mycophenolate mofetil hydrochloride (IV), mycophenolate sodium (PO), methotrexate, tacrolimus, sirolimus, thalidomide, leflunomide, mizoribine, ciclosporin). Intravenous immunoglobulin (IVIG). Plasmapheresis, leukapheresis, Time Period: 90 days; Therapy: A non-biologic investigational agent (i.e. not approved for sale in the country in which it is being used). Intravenous corticosteroid, Adrenocorticotropic hormone (ACTH). Aliskiren. A change in dose of >50% for angiotensin pathway antihypertensive (e.g., ACE inhibitor, angiotensin receptor blocker), Time Period: 60 days; Therapy: A live vaccine. Greater than 30mg/day corticosteroid, Time Period: 30 days; Therapy: Greater than 10mg/day corticosteroid. A change in dose of a corticosteroid. Note: Changes to inhaled steroids and new topical immunosuppressive agents (e.g., eye drops, topical creams) are allowed, Time Period: 14 days.
* Transplantation: Have a history of a major organ transplant (e.g., heart, lung, kidney, liver) or hematopoietic stem cell/marrow transplant.
* Cancer: Have a history of malignant neoplasm within the last 5 years, except for adequately treated cancers of the skin (basal or squamous cell) or carcinoma in situ of the uterine cervix.
* Acute or chronic infection: Have required management of acute or chronic infections such as currently on any suppressive therapy for a chronic infection such as tuberculosis, pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster and atypical mycobacteria); or hospitalisation for treatment of infection within 60 days prior to Day 0; or use of parenteral (IV or IM) antibiotics (anti-bacterials, anti-virals, anti-fungals, or anti-parasitic agents) within 60 days prior to Day 0.
* Liver disease: Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Other diseases/conditions: Have clinical evidence of significant unstable or uncontrolled acute or chronic diseases not due to IMN (i.e., cardiovascular, pulmonary, haematologic, gastrointestinal, hepatic, renal, neurological, malignancy or infectious diseases) which, in the opinion of the investigator, could confound the results of the study or put the subject at undue risk; or have a planned surgical procedure or a history of any other medical disease (e.g. cardiopulmonary), laboratory abnormality, or condition (e.g., poor venous access) that, in the opinion of the investigator, makes the subject unsuitable for the study.
* Positive serology: Have a historically positive HIV test or test positive at screening for HIV. Serologic evidence of Hepatitis B (HB) infection based on the results of testing for HBsAg, anti-HBc and anti-HBs. Positive test for Hepatitis C antibody confirmed on the same sample with a Hepatitis C RIBA immunoblot assay if available.
* Liver function tests: Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) >=2x upper limit of normal (ULN); alkaline phosphatase and bilirubin >1.5xULN (isolated bilirubin >1.5ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Immunodeficiency: Have an IgA deficiency (IgA level < 10 mg/dL) or have IgG level <250 mg/dL and have previously received any non-glucocorticoid immunosuppression during the previous 6 months.
* Laboratory test abnormalities: Have clinically significant abnormalities in screening laboratory assessments (not related to the disease), as judged by investigator.
* Drug sensitivity / Anaphylaxis: History of sensitivity or intolerance to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation. History of an anaphylactic reaction to parenteral administration of contrast agents, human or murine proteins or monoclonal antibodies.
* Suicidality: Subjects who have evidence of serious suicide risk including any history of suicidal behaviour in the last 6 months and/or any suicide ideation of type 4 or 5 on the Columbia Suicide-Severity Rating Scale (C-SSRS) in the last 2 months or who in the investigator's judgement, pose a significant suicide risk.
* Substance abuse: Evidence of current drug or alcohol abuse or dependence.
* Blood donation: Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of remission (complete [CR] or partial [PR]) at Week (WK) 104 | 104 weeks
  CR: urine protein to creatinine ratio (uPCR) <30 mg/mmol (proteinuria <0.3 g/24 hr) with no worsening of renal function (<15% estimated glomerular filtration rate [eGFR] reduction from baseline [BL]).PR: uPCR <350 mg/mmol (proteinuria <3.5g/24 hrs) but >=30 mg/mmol (proteinuria >=0.3g/24 hrs) AND a decrease of >50% from BL based on uPCR, with no worsening of renal function. uPCR: Mean from 2 consecutive 24 hr urine collections (pre and post dose or pre and post visit). eGFR: BL will be defined as mean of screening and Day 0 values. For WK 104 assessment, will be analysed at both WK 100 and 104

SECONDARY OUTCOMES:
Incidence of progression of IMN or failure to respond | Upto Week 104
  Defined by at least one of the following:1.Persistent symptomatic nephrotic syndrome potentially necessitating rescue therapy 2.End Stage Renal Disease (eGFR <15 mL/min/1.73m^2,dialysis or transplantation).3.Clinical thromboembolic events. 4.Death
Time to complete remission | Up to Week 104
  Complete Remission (CR) is defined as uPCR <30 mg/mmol (proteinuria <0.3 g/24 hrs) with no worsening of renal function (less than 15% reduction in estimated eGFR from baseline)
Time to partial remission | Up to Week 104
  Partial Remission (PR) is defined as uPCR <350 mg/mmol (proteinuria <3.5 g/24 hrs) but >=30 mg/mmol (proteinuria >=0.3g/24 hrs) AND a decrease of >50% from baseline (Day 0) based on uPCR, together with no worsening of renal function (less than 15% reduction in eGFR from baseline)
Change from baseline in proteinuria levels at Week 104 | Week 0 and Week 104
  Mean uPCR from 2 consecutive 24 hr urine collections (pre and post dose or pre and post visit)
Change from baseline in serum albumin levels at Week 104 | Week 0 and Week 104
  Albumin levels will be measured to determine hypoalbuminaemia. Baseline will be defined as mean of screening and Day 0 values. For the week 104 assessment, albumin will be analyzed at both weeks 100 and 104.
Change from baseline in eGFR at Week 104 | Week 0 and Week 104
  Baseline will be defined as mean of screening and Day 0 values. For the week 104 assessment, eGFR will be analyzed at both weeks 100 and 104.
Time to first thromboembolic event | Up to Week 104
  Thromboembolism is a formation in a blood vessel of a clot (thrombus) that breaks loose and is carried by the blood stream to plug another vessel. Thromboembolic event is a complication of nephrotic syndrome.
Change from baseline in KDQOL-36 score at Week 104 | Week 0 and Week 104
  The Kidney Disease Quality of Life (KDQOL- 36) consists of the SF-12 Physical Health and Mental Health Composite scores along with the Burden of Kidney Disease and Effects of Kidney Disease subscales.
Incidence of partial remission at Week 104 | Week 104
  Partial Remission (PR) is defined as uPCR <350 mg/mmol (proteinuria <3.5g/24 hrs) but >=30 mg/mmol (proteinuria >=0.3 g/24 hrs) AND a decrease of >50% from baseline (Day 0) based on uPCR, together with no worsening of renal function (less than 15% reduction in eGFR from baseline)
Incidence of complete remission at Week 104 | Week 104
  Complete Remission (CR) is defined as uPCR <30 mg/mmol (proteinuria <0.3 g/24 hrs) with no worsening of renal function (less than 15% reduction in estimated eGFR from baseline)
Duration of remission (complete or partial) | Up to Week 104
  The duration of remission (complete or partial) will be assessed to evaluate length of effect of belimumab.
Risk-benefit calculation based on key efficacy and safety endpoints using a clinical utility index | Up to Week 104
  A clinical utility index will be developed to objectively measure benefit over standard practice in a quantitative manner.
Incidence of serious adverse events (SAEs) | Up to Week 104
  SAEs are medical occurrences not due to the disease (unless more severe than expected), but which result in death, disability, incapacity, are life threatening, require or prolong hospitalization, are associated with specified liver injury/impaired function and other defined criteria. SAEs beyond Week 104 will be assessed as 'Other endpoints' or 'Long Term Follow-up endpoints'
Incidence of adverse events (AEs) of special interest | Up to Week 104
  AEs of special interest will include: Serious infusion reactions/hypersensitivity/anaphylaxis, fatal events; serious malignancies; serious infections including herpes zoster; cardiovascular SAEs (fatal and non-fatal events) including arrhythmia, congestive heart failure, cerebrovascular accident, deep vein thrombosis, myocardial infarction/unstable angina, peripheral arterial thromboembolism, revascularization; SAEs suggestive of suicidal or self-harming behavior
Safety assessed by evaluation of Adverse events, clinical laboratory assessments, vital signs and immunogenicity | Up to 116 Weeks
  Safety and tolerability assessed by evaluation of adverse events (AE), clinical laboratory assessments (clinical chemistry, haematology and urinalysis), vital signs and immunogenicity. Including infusion-related and hypersensitivity reactions, infections and malignancies
Survival without renal progression | From start of treatment up to 7 years
  Subjects will be followed annually for 5 years after Week 104 in the main clinical study or until ESRD or death, whichever is earlier for analysis of survival without renal progression. Survival without renal progression will be defined as the time from start of treatment until decrease in eGFR from baseline at entry into the study by greater than 20% OR end stage renal disease (eGFR <15 mL/min/1.73 m^2, start of dialysis or renal transplantation) OR death.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (29):
- United States (2):
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Chapel Hill, North Carolina
- GSK Investigational Site, New Lambton, New South Wales, Australia
- Canada (2):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, London, Ontario
- GSK Investigational Site, Prague, Czechia
- France (4):
  - GSK Investigational Site, Amiens
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Toulouse
- Germany (7):
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Aachen, North Rhine-Westphalia
  - GSK Investigational Site, Solingen, North Rhine-Westphalia
  - GSK Investigational Site, Berlin, State of Berlin
- Italy (2):
  - GSK Investigational Site, Lecco, Lombardy
  - GSK Investigational Site, Lido Di Camaiore (LU), Tuscany
- Netherlands (2):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Nijmegen
- Spain (3):
  - GSK Investigational Site, L'Hospitalet de Llobregat
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Valencia
- United Kingdom (5):
  - GSK Investigational Site, Cardiff
  - GSK Investigational Site, Gloucester
  - GSK Investigational Site, Leicester
  - GSK Investigational Site, London
  - GSK Investigational Site, Reading

REFERENCES:
- [Derived] von Groote TC, Williams G, Au EH, Chen Y, Mathew AT, Hodson EM, Tunnicliffe DJ. Immunosuppressive treatment for primary membranous nephropathy in adults with nephrotic syndrome. Cochrane Database Syst Rev. 2021 Nov 15;11(11):CD004293. doi: 10.1002/14651858.CD004293.pub4. PMID 34778952